CLINICAL TRIAL: NCT00005632
Title: Vaccination of Prostate Cancer Patients With MUC-1-KLH Conjugate Plus the Immunological Adjuvant QS21: A Trial Examining the Immunogenicity of MUC-1 Glycopeptide Conjugate
Brief Title: Vaccine Therapy Plus QS21 in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-040; MSKCC-99040; NCI-G00-1773
Record Dates: First submitted 2000-05-02; First posted 2004-07-19 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Vaccine (Experimental): Patients sequentially will receive glycosylated MUC-1-KLH vaccines at 3ug per vaccination.
  Interventions: Biological: MUC1-KLH vaccine/QS21

INTERVENTIONS:
Biological: MUC1-KLH vaccine/QS21

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Combining a vaccine with QS21 may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy plus immune adjuvant QS21 in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if immunization with glycosylated MUC-1 antigen containing MUC-1 (106) with keyhole limpet hemocyanin conjugate plus immunological adjuvant QS21 induces an antibody, helper T cell and/or cytotoxic T cell response against MUC-1 in patients with prostate cancer expressing MUC-1. II. Determine post-immunization changes in PSA levels and other objective parameters or disease (radionuclide bone scan and/or measurable disease if present) in these patients after receiving this therapy.

OUTLINE: Patients receive glycosylated MUC-1 antigen containing MUC-1 (106) with keyhole limpet hemocyanin conjugate subcutaneously (SQ) plus immunological adjuvant QS21 SQ on weeks 1-3, 7, 15, and 27 for a total of 6 vaccinations. Patients are followed every 3 months for 1 year or until documented disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed prostate cancer No radiographic evidence of metastatic disease Must show signs of disease progression 3 or more rising PSA values documented, taken at no less than weekly intervals, to greater than 50% above baseline PSA PSA at least 1.0 ng/mL (post prostatectomy) OR 2.0 ng/mL (post radiation) Evaluable disease by serial changes in PSA Progression after primary therapy to include surgery or radiotherapy (with or without neoadjuvant androgen ablation), or intermittent hormonal therapy with noncastrate levels of testosterone (greater than 50 ng/mL) allowed No soft tissue and/or bone disease or androgen independent disease with no evidence of radiographic disease No symptomatic disease or anticipated to be symptomatic within 6 months No active CNS or epidural tumor

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 6 months Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL OR SGOT less than 3 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No New York Heart Association class III-IV heart disease Pulmonary: No severe debilitating pulmonary disease Other: No other malignancy within past 5 years except nonmelanoma skin cancer No concurrent infection requiring antibiotics No narcotic dependent pain No positive stool guaiac excluding hemorrhoids No history of documented radiation induced proctitis No allergy to seafood

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior murine monoclonal antibody therapy No other concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 2 weeks since prior changes in hormonal therapy including prednisone or dexamethasone At least 8 weeks since prior suramin OR documented plasma concentration less than 50 mg/mL (replacement doses of hydrocortisone allowed) Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy to only measurable lesion Surgery: See Disease Characteristics No concurrent surgery Other: No other concurrent anticancer agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1999-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States